CLINICAL TRIAL: NCT03549026
Title: Analgesic Efficacy of Duloxetine in Patients Undergoing Lumbar Discectomy: Randomized Trial
Brief Title: Analgesic Efficacy of Duloxetine in Patients Undergoing Lumbar Discectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, lecturer of anesthesia and pain management , Assuit university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0006563-535
Record Dates: First submitted 2018-05-20; First posted 2018-06-07 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- duloxitine group (Experimental): Patients will receive single oral dose of duloxetine capsule, 60 mg, 2 hours before operation and will be anesthetized with general anesthesia that includes, Induction of anesthesia will be done by intravenous fentanyl, 2 µg / kg and propofol 1 - 2 mg / kg. Endotracheal intubation will be achieved by cis-atracurium, 0.15 mg / kg. Maintenance of anesthesia will be done by isoflurane and cis-atracurium, 0.03 mg / kg on demand. Additional intraoperative analgesia will be consisted of administration of intravenous boluses of fentanyl, 50 µg according to the attending anesthesiologist's decision. At the end of surgery, muscle relaxation was reversed using neostigmine 0.05 mg / kg and atropine 0.01 mg / kg.
  Interventions: Drug: Duloxetine
- placebo group (Placebo Comparator): Patients will receive single oral dose of placebo capsule, 2 hours before operation and will be anesthetized with general anesthesia that includes, Induction of anesthesia will be done by intravenous fentanyl, 2 µg / kg and propofol 1 - 2 mg / kg. Endotracheal intubation will be achieved by cis-atracurium, 0.15 mg / kg. Maintenance of anesthesia will be done by isoflurane and cis-atracurium, 0.03 mg / kg on demand. Additional intraoperative analgesia will be consisted of administration of intravenous boluses of fentanyl, 50 µg according to the attending anesthesiologist's decision. At the end of surgery, muscle relaxation was reversed using neostigmine 0.05 mg / kg and atropine 0.01 mg / kg.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Duloxetine — The investigator will give the patients duloxetine capsule 60 mg orally before operation (skin incision) and anesthetize them with general anesthesia, then the investigator will test the postoperative analgesic efficacy in the form of 24 h analgesic consumption
  Arms: duloxitine group
Drug: placebo — Patients will receive single oral dose of placebo capsule, 2 hours before operation and will be anesthetized with general anesthesia that includes, Induction of anesthesia will be done by intravenous fentanyl, 2 µg / kg and propofol 1 - 2 mg / kg. Endotracheal intubation will be achieved by cis-atracurium, 0.15 mg / kg. Maintenance of anesthesia will be done by isoflurane and cis-atracurium, 0.03 mg / kg on demand. Additional intraoperative analgesia will be consisted of administration of intravenous boluses of fentanyl, 50 µg according to the attending anesthesiologist's decision. At the end of surgery, muscle relaxation was reversed using neostigmine 0.05 mg / kg and atropine 0.01 mg / kg
  Arms: placebo group

SUMMARY:
Duloxetine is a serotonin-norepinephrine reuptake inhibitor primarily used for treatment of major depression and anxiety. Duloxetine also has been used in the treatment of chronic pain conditions, such as osteoarthritis and musculoskeletal pain. There are few studies examining its effect for acute pain. The objective of this study is to evaluate the analgesic effect of duloxetine for patients undergoing lumbar discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar discectomy

Exclusion Criteria:

* Patients on regular opioid therapy
* Uncontrolled hypertensive patients
* Patients with ischemic heart disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-25 (Estimated)

PRIMARY OUTCOMES:
the first 24 hour morphine consumption | the first postoperative 24 hour
  the first 24 hours cumulative morphine consumed by the patient via patient controlled analgesic device (PCA), set to deliver 2 mg morphine bolus with lockout interval 15 min, without background infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt